# Informed Consent Form

Study Title: Erectile Dysfunction and the Mind: Evaluating the Influence of Depression and

Illness Beliefs on Treatment Progression

NCT Number: NCT06996925

Principal Investigator: Dr. Nazım Furkan Günay

Institution: Haseki Training and Research Hospital

Document Date: August 6, 2025

Email: nfurkangunay@gmail.com

#### Introduction

You are invited to participate in a clinical study titled "Erectile Dysfunction and the Mind: Evaluating the Influence of Depression and Illness Beliefs on Treatment Progression." Before you decide, it is important that you understand why this research is being conducted and what your participation will involve.

## **Purpose of the Study**

This study aims to investigate the psychological and emotional aspects of erectile dysfunction, specifically how patients' beliefs about their illness and their emotional state, including depression, affect their overall well-being and treatment outcomes.

#### **Duration and Procedures**

You will be asked to attend two visits:

- 1. At the first visit, you will be asked to complete three brief questionnaires regarding:
  - Your erectile function (IIEF-5),
  - Your emotional state (PHQ-9),
  - Your thoughts and beliefs about your condition (B-IPQ).
- 2. One month later, you will complete the same questionnaires again.

There are no medical treatments or interventions involved in this study.

## **Benefits of Participation**

Although there may be no direct benefit to you, your participation will help us better understand the impact of psychological factors on erectile dysfunction. The findings may improve how care is provided to future patients facing similar challenges.

#### **Risks and Discomforts**

There are no physical risks in this study. However, some questions in the surveys may evoke emotional discomfort. You may skip any question you do not wish to answer or withdraw from the study at any time without penalty.

## **Confidentiality**

All information you provide will remain strictly confidential and will only be used for research purposes. Your identity will not be revealed in any reports or publications resulting from this study.

## **Voluntary Participation**

Your participation is entirely voluntary. You may refuse to participate or withdraw from the study at any point without giving any reason. Your decision will not affect your medical care in any way.

# **Questions and Contact Information**

If you have any questions about the study or wish to withdraw your participation, please contact: Dr. Nazım Furkan Günay

Email: nfurkangunay@gmail.com

#### Consent Statement

I have read and understood the information provided above. I have had the opportunity to ask questions and have received satisfactory answers. I understand that my participation is voluntary and that I may withdraw at any time. I freely agree to take part in this study.

| Participant Name and Surname: _ |
|---------------------------------|
| Signature: |
| Date: |
| Researcher Name and Surname: |
| Signature: |

| Date: |
|-------|
|-------|